CLINICAL TRIAL: NCT05615714
Title: Paresthesia-free Peripheral Nerve Field Stimulation for Trigeminal Neuralgia: a Double-blinded, Randomized Trial (FreeST Trial)
Brief Title: Paresthesia-free Peripheral Nerve Field Stimulation for Trigeminal Neuralgia (FreeST Trial)
Acronym: FreeST
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Mojgan Hodaie, Professor, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 21-6219
Record Dates: First submitted 2022-10-30; First posted 2022-11-14 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Trigeminal Neuralgia; Facial Pain
Keywords: Peripheral Nerve Field Stimulation
MeSH Terms: conditions — Trigeminal Neuralgia; Facial Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paresthesia-Free Stimulation (Experimental): Duration: 2 weeks
  Interventions: Other: Paresthesia-free Peripheral Nerve Field Stimulation
- Sham Stimulation (Sham Comparator): Duration: 2 weeks
  Interventions: Other: Sham stimulation

INTERVENTIONS:
Other: Paresthesia-free Peripheral Nerve Field Stimulation — High frequency and sub-paresthesia threshold intensity parameters will be used for paresthesia-free stimulation of trigeminal nerve branches.
  Arms: Paresthesia-Free Stimulation
Other: Sham stimulation — Stimulation will be turned off.
  Arms: Sham Stimulation

SUMMARY:
Study type: Prospective, double-blinded, double arm, cross-over, randomized controlled clinical trial.

Brief protocol:

Postoperative week 0-2 -> Conventional parameters (parameters tested during trial period)

Postoperative week 2-6 -> Sham stimulation (2 weeks) and paresthesia-free stimulation (2 weeks) double-blind crossover design

Postoperative week 6 - month 12 -> Parameters that patients feel more benefit from

DETAILED DESCRIPTION:
Background:

Peripheral Nerve Field Stimulation (PNFS) has been utilized for the treatment of facial pain for around 60 years, and the commercial devices needed to deliver PNFS have been available for around 30 years. The safety and efficacy of the procedure has been demonstrated by various uncontrolled observational studies. It serves as a part of daily neurosurgical practice for selected patients in UHN Toronto Western Hospital. This therapeutic modality involves subcutaneous implantation of electrodes in the vicinity of trigeminal nerve branches and application of electrical current using a permanently implanted pulse generator (IPG). Similar to other forms of neuromodulation, PNFS is non-ablative, reversible, adjustable and associated with a relatively low risk of severe complications. A meta-analysis of paresthesia-inducing (PI) PFNS studies in the literature revealed a treatment efficacy of 75% decrease in VAS scores (mean difference: -6.32 out of 10) with PNFS utilization for facial pain. (PMID: 35180702)

Study design:

Patients who underwent a successful unilateral PNFS implantation surgery (trial and permanent implantation) for a facial pain syndrome as a standard of care treatment, will be screened for inclusion after permanent implantable pulse generator (IPG) implantation. Upon consent, the investigators will set up participants' IPG to deliver stimulation with parameters tested during the trial period (paresthesia-inducing parameters) for 2 weeks. The participants will come back to hospital at postoperative week 2 and will be randomized (1:1 ratio) between the two arms of the study (Group 1= sham, Group 2= paresthesia-free (PF) stimulation). Each participant will consecutively experience all two stimulation groups by 2-week periods in a crossover design. Both participants and clinical investigators that will assess the pain will be blind during the study period (between postoperative week 2 and 6). After 6 weeks, the treatment arms will be merged and all the participants will receive any stimulation parameter that they feel more benefit from ("best" parameter). Outcomes will be assessed 6 and 12 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a medically-refractory unilateral facial pain syndrome as defined by the Burchiel classification but excluding atypical facial pain (somatoform pain disorder)
* Recent successful PNFS trial and permanent implantation surgery
* Average preoperative episodic/constant pain intensity of 5 or greater out of 10 cm on the VAS
* Capable of providing informed consent and complying with study procedures
* Patients may or may not use a pain medication at the time of recruitment. Medications allowed during the study are long-acting/modulatory analgesics (anticonvulsants such as carbamezapine, oxcarbazepine, pregabalin, gabapentin, lamotrigine; baclofen, botox injections) and short-acting analgesics (non-steroid anti-inflammatory drugs, short-acting opioids, lidocaine or sumatriptan injections)

Exclusion Criteria:

* Currently in a clinical trial involving an investigational product or non-approved use of a drug or device.
* Active psychiatric disorder or other known condition that can significantly impact pain perception
* Patients with a revision surgery of a PNFS system by any reason (history of trigeminal pain surgery of other types (i.e., microvascular decompression, gamma knife, percutaneous rhizotomies) are not exclusion criteria)
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-10-28 (Estimated); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Score Change | Postoperative week 2 to week 6
  VAS score change between sham condition (postop week 2-4 or postop week 4-6) and Paresthesia-free stimulation condition (postop week 2-4 or postop week 4-6) VAS score ranges from 0 to 100 mm (or 0 to 10 cm). Higher score is worse outcome.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Score Change | Postoperative week 0 to week 6
  Score changes between sham condition (postop week 2-4 or postop week 4-6), Paresthesia-free stimulation condition (postop week 2-4 or postop week 4-6) and Paresthesia-inducing stimulation condition (postop week 0-2) Non-independent within-group comparison VAS score ranges from 0 to 100 mm (or 0 to 10 cm). Higher score is worse outcome.
Barrow Neurological Institute (BNI) pain intensity score change | Postoperative week 0 to week 6
  Score changes between sham condition (postop week 2-4 or postop week 4-6), Paresthesia-free stimulation condition (postop week 2-4 or postop week 4-6) and Paresthesia-inducing stimulation condition (postop week 0-2) Non-independent within-group comparison BNI score ranges from 1 to 5. Higher score is worse outcome.
Brief Pain Inventory (BPI) score change | Postoperative week 0 to week 6
  Score changes between sham condition (postop week 2-4 or postop week 4-6), Paresthesia-free stimulation condition (postop week 2-4 or postop week 4-6) and Paresthesia-inducing stimulation condition (postop week 0-2) Non-independent within-group comparison BPI-Pain Severity Score and BPI-Pain Interference Score range from 0 to 10. Higher score is worse outcome.
Clinician and Patient Global Impression of Change Scale and Patient satisfaction scale score change | Postoperative week 0 to week 6
  Score changes between sham condition (postop week 2-4 or postop week 4-6), Paresthesia-free stimulation condition (postop week 2-4 or postop week 4-6) and Paresthesia-inducing stimulation condition (postop week 0-2) Non-independent within-group comparison Clinician and Patient Global Impression of Change Scale (range from 1 to 7) and Patient satisfaction scale (range from 1 to 5). Higher score is worse outcome.
Adverse effect Profile | Postoperative week 0 to month 12
  Adverse effect Profile
Ratio of patients who chose paresthesia-free or paresthesia-inducing stimulation at week 6, month 6 and 12 | Postoperative week 6, month 6 and 12
  paresthesia-free or paresthesia-inducing stimulation
fMRI BOLD signal change | Between postoperative month 6 and 12
  IPG ON>OFF BOLD signal change (both paresthesia-free and Paresthesia-inducing conditions will be tested)
Visual Analogue Scale (VAS) Score Change | Postoperative month 6 and 12
  Score changes between baseline and postoperative 6 and 12 months VAS score ranges from 0 to 100 mm (or 0 to 10 cm). Higher score is worse outcome.
Barrow Neurological Institute (BNI) pain intensity score change | Postoperative month 6 and 12
  Score changes between baseline and postoperative 6 and 12 months BNI score ranges from 1 to 5. Higher score is worse outcome.
Brief Pain Inventory (BPI) score change | Postoperative month 6 and 12
  Score changes between baseline and postoperative 6 and 12 months BPI-Pain Severity Score and BPI-Pain Interference Score range from 0 to 10. Higher score is worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mojgan Hodaie, MD, MSc, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec